CLINICAL TRIAL: NCT02605785
Title: A Molecular Anatomic Imaging Analysis of Tau in Progressive Supranuclear Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Keith A. Josephs, Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-004618
Record Dates: First submitted 2015-11-03; First posted 2015-11-16 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Progressive Supranuclear Palsy
Keywords: PSP
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tau PET Scan, F-18 AV 1451 (Experimental): All subjects will received a Tau PET scan.
  Interventions: Drug: F-18 AV 1451

INTERVENTIONS:
Drug: F-18 AV 1451 — Tau PET scan
  Other Names: Tau binding agent

SUMMARY:
This study is designed to learn more about overall tau burden in the brain of patients with Progressive Supranuclear Palsy (PSP).

ELIGIBILITY:
Inclusion Criteria:

* Must be over 35 years of age and present with gradual progression of PSP-related symtoms
* Must have an informant or study partner that can provide independent information of functioning.
* Must meet criteria for possible or probable Progressive Supranuclear Palsy. To fulfill criteria for possible PSP, subjects must have a gradually progressive disorder with either vertical (upward or downward) supranuclear palsy or both slowing of vertical saccades and prominent postural instability with falls in the first year of disease onset. To fulfill criteria for probable PSP, subjects must have vertical (upward or downward gaze) supranuclear palsy and prominent postural instability with falls in the first year of disease onset.

Exclusion Criteria:

* Subjects will be excluded if they meet criteria for another neurodegenerative disease (including corticobasal syndrome, frontotemporal dementia, primary progressive aphasia, Alzheimer's disease, multiple system atrophy and Parkinson's disease) or do not have the symptoms necessary to fulfill inclusion criteria for possible PSP.
* Subjects with concurrent illnesses that could account for their symptoms, such as traumatic brain injury, encephalitis, strokes or developmental syndromes will be excluded.
* Women that are pregnant or post-partum and breast-feeding will be excluded.
* Subjects will be excluded from the study if they have any of the following genetic conditions which can increase the chance of cancer: Cowden disease, Lynch syndrome, hypogammaglobulinemia, Wiskott-Aldrich syndrome, and Down's syndrome.
* Subjects will also be excluded if MRI is contraindicated (metal in head, cardiac pace maker, e.t.c.), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma, intracranial neoplasm or large cortical infarcts), or if they are medically unstable or are on medications that might affect brain structure or metabolism (e.g. chemotherapy).
* Subjects will also be excluded if they do not have an informant, or do not consent to research.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2015-11; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The investigators will be looking at the amount of Tau protein in the brain of patients with PSP. | 5 years

SECONDARY OUTCOMES:
Rates of change in tau-PET burden over time. | baseline, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whitwell, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials